# **CLINICAL TRAIL PROTOCOL**

Protocol Title: Immunogenicity and Safety of Quadrivalent Influenza Vaccine In 6 to 35 months population: a Randomized, Double-blind, Parallel-group II phase of clinical trials

Collaborators: Henan Center for Disease Control and Prevention

Sponsor: Shanghai Institute of Biological Products

Document Date: January 1, 2020

#### BACKGROUD INFORMATION

Since 1978, influenza A (H1N1) influenza A (H3N2) and influenza B virus are commonly circling every season. Then, the trivalent influenza vaccine had been developed against the three kinds of influenza virus (H1N1 and H3N2 and B). According to the result of global influenza surveillance, the World Health Organization has been to predict the next season's pandemic strains for more than 30 years. WHO recommended vaccine components containing two subtypes of A influenza virus (H1N1 and H3N2) and a subtype of B influenza virus (B/Victoria lineage or B/Yamagata lineage). However, since the 2001-2002 influenza season, two strains of influenza B have been circulating together. This made it difficult to predict the dominant strain of influenza B in the next influenza season. Several studies demonstrated that in 7 of the past 13 seasons, major cycling subtype of B virus strains was not included in the vaccine, which significantly reduces the immunological effects of the influenza vaccine. Unincluded subtype B influenza virus caused a potential threat to human beings. To expand the broad protection of the seasonal influenza vaccine and improve the protective effect of the vaccine, many influenza vaccine manufacturers had actively carried out the development of the quadrivalent influenza vaccine, which has become an important direction for the upgrading of influenza vaccine.

At the same time, several studies showed that the influenza vaccine induces a poor immune response in young children. Unvaccinated children below 3 years older were induced by vaccine weaker than unvaccinated children above 3 years older younger or vaccinated children below 3 years older, especially for the B subtype influenza virus. For 6 ~ 35 months old children were recommended vaccination dosage of 0.25 ml antigen of influenza inactivated vaccines. This recommendation was based on the observation in the 1970s of increased adverse reactivity in younger children with an adult's dosage of whole-virus inactivated influenza vaccines, especially the fever but at present in the seasonal flu vaccine has been without the use of an inactivated virus. The safety and immunogenicity of 0.5ml and 0.25ml dosage antigen of vaccine were evaluated in 6~35 months children in a large number of clinical trials. The results showed that the high dosage of the split vaccine was well tolerated and could induce a strong immune response. Hence, in 2016, the FDA approved the adult dosage of the influenza vaccine for children above 6 months. Besides, many countries such as Canada, Brazil, Mexico, Finland, and Britain approved dosage of 15ug and

7.5 µg antigen for children below 3 years.

Given the situation of children-using the influenza vaccine, we carried out the clinical trial of the quadrivalent influenza vaccine suitable for children aged 6 to 35 months, which is of great significance for children to prevent influenza in China.

#### **STUDY OBJECT**

To evaluate the immunogenicity and safety of 2 doses of quadrivalent influenza virus split vaccine (0.25ml/ dose and 0.5ml/ dose) in healthy population aged 6-35 month., so as to provide a data support for phase III clinical trials.

#### STUDY DESIGN

A randomized, double-blind, parallel control design was set to enroll 1,980 healthy subjects aged 6-35 months. Subjects were randomly inoculated with experimental vaccine 1, experimental vaccine 2, control vaccine 1 or control vaccine 2 in a ratio of 2:2:1:1 for safety and immunogenicity evaluation. The inoculation time was 0 and 28 days.

#### Immunogenicity observation

- All subjects were required to take bloody samples for 2 times, each time about 3.0ml, for the detection of influenza virus HI antibody:
- First time: before the first dose;
- Second dose: 28 (+10) days after the second dose.
- After 30 days of safety observation and 28 days of immunogenicity test results after 2 doses of immunization, uncovered blind and the immunogenicity results were statistically analyzed.

#### Safety observation:

 All adverse events were collected at 0-7 days after immunization, all adverse events at 0-28/30 days, and all serious adverse events (SAE) within 6 months (180 days) after 2 doses of vaccine immunization.

| | | | | Inoculation | Serum | |
|---|---|---|---|---|---|---|
| Age | Group | Vaccine | Number | | collection | Safety observation |
| | | | | (uay) | (day) | |

| | | | | | | 1. Adverse events within |
|---|---|---|---|---|---|---|
| | A1 | Experimental Vaccine 1 | 660 | | | 28/30 days after each |
| | | | | | | dose of immunization |
| | A2 | Experimental Vaccine 2 | 330 | | | were collected; |
| 6-35 | | • | | 0, 28 | 0, 56 | 2. Serious adverse events |
| Month | B1 | Control Vaccine 1 | | (+10) | (+10) | (SAE) were collected |
| | | | 330 | | | within 6 months after the |
| | | | | | | first dose of inoculation |
| | B2 | Control Vaccine 2 | 660 | | | and after the whole |
| | | | | | | course of immunization. |
| Total | | | 1980 | | | |

#### STUDY ENDPOINT

#### Immunogenicity

- (1) 28 days after receiving two doses of vaccine in subjects aged 6-35 months, seroconversion rate of HI antibodies against any subtype of influenza virus in each group.
- (2) 28 days after receiving two doses of vaccine in subjects aged 6-35 months, seroprotection rate of HI antibodies against any subtype of influenza virus in each group.
- (3) 28 days after receiving two doses of vaccine in subjects aged 6-35 months, GMT and GMI of HI antibodies against any subtype of influenza virus in each group.

#### Safety

- (1) The proportion of all adverse reactions/events in each group through 30 days after the second dose.
- (2) The proportion of serious adverse events (SAE) within 6 months after inoculation in each group.

## **SAFETY OBSERVATION**

Systemic adverse reactions: Fever, Diarrhea, constipation, difficulty swallowing, anorexia, vomiting, nausea, muscle pain (not the vaccination site), arthritis, joint pain, headache, new convulsions, cough and difficulty breathing, the vaccination site itching (no skin damage), abnormal skin and mucosa, insomnia, irritability, or inhibiting, acute allergic reaction to pain, fatigue, lack of power, not the vaccination site.

Local adverse reactions: pain, induration, swelling, rash, redness, itching

IMMUNOGENICITY OBSERVATION

Seroconversion: 1:10 is the lowest serum dilution. Prevaccination HI titer < 1:10 and

postvaccination titer  $\geq 1:40$  or a prevaccination titer  $\geq 1:10$  and at least a 4-fold increase in the

postvaccination titer

Seroprotection: Postvaccination titer  $\geq 1:40$  is considered to have antibody protection.

GMT: geometric mean titer.

GMI: GMT increase fold.

**EVALUATION CRITERIA OF SAFETY** 

The safety evaluation of each group will be divided into three stages. From the first dose

inoculation to day 7 after inoculation; From the first dose inoculation to day 21 after inoculation;

From the second dose inoculation to day 30 after the second dose inoculation. The first stage is the

basis for the follow-up group of the same vaccine, and will be carried out under blind. The latter

two stages are the basis for evaluation of vaccine safety, and will be carried out under unblind. If each evaluation is not found level 4 local and systemic adverse reactions associated with vaccine

and the total incidence rate of level 3 of local and systemic adverse reactions and abnormal

laboratory test which associated with the vaccination is lower than 15%, that the vaccine will be

acceptable safety.

**EVALUATION CRITERIA OF IMMUNOGENICITY** 

If seroconversion rate is higher than 40%, the antibody protection rate higher than 70%, GMI

more than 2.5 times, the vaccine will be acceptable immunogenicity.

**STUDY STATUS** 

Record Verification: January 2020

Study Start: April 2020

Primary Completion: August 2020

Study Completion: March 2021

**ELIGIBILITY** 

Inclusion Criteria

Healthy infants aged 6-35 months.

Volunteer legal guardian or client informed consent, voluntarily participate in and sign informed consent.

The volunteer legal guardian or client has the ability (non-illiterate) to understand the study procedures, to use a thermometer, scale, and fill in a diary card as required, and be able to complete the clinical study in compliance with the clinical trial protocol.

#### **Exclusion Criteria**

The underarm body temperature on the day of enrollment was > 37.0°C.

Have been suffering from influenza within the previous 3 months (confirmed by either clinical, serological or microbiological methods).

Any previous influenza vaccination (registered or experimental) within 6 months or any planned influenza vaccination during the study period.

Allergic to any component of the vaccine, a history of allergic reactions to eggs or gentamicin sulfate.

A history of severe allergy to any vaccine or drug.

Preterm birth (delivered before 37 weeks of gestation), low birth weight baby (birth weight < 2300g for girls, <2500g for boys).

Dystocia, asphyxia rescue, nervous system damage history;

Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.

Acute illness, severe chronic illness or acute attack of chronic disease on the day of vaccination;

A history of live attenuated vaccination within 14 days prior to vaccination and a history of other vaccinations within 7 days prior to vaccination;

Patients who received immunoenhancement or inhibitor therapy within 3 months (continued oral or intravenous administration for more than 14 days);

Congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;

History of asthma, past two years of instability requiring emergency treatment, hospitalization, intubation, oral or intravenous administration of corticosteroids;

Have received blood or blood-related products;

A history of convulsion, epilepsy, encephalopathy, guillain-barre syndrome, a history of mental illness or a family history;

A history of abnormal coagulation function (such as coagulation factor deficiency,

coagulation disease);

Planning to relocate before the end of the study or to leave for an extended period during the scheduled study visit;

Participating in or planning to participate in other clinical trials in the near future;

The investigators determined that any conditions were inappropriate to participate in the clinical trial.

#### **DATA STATISTICS**

#### Statistics analysis of immunogenicity

The prevaccination and postvaccination geometric mean of antibody and its 95% confidence interval (confidence interval, CI) will be described. The postvaccination serum conversion rate and protection rate of antibody and their 95% CI will be described.

Comparisons will be conducted to evaluate differences in response between study groups using a  $\chi^2$  test or Fisher's exact test to compare to the difference of serum conversion rate and protection rate. Statistical significance will be considered at a level of  $\alpha$  = 0.05 and all tests will be 2-sided.

If serum HI antibody conversion rate is more than 40%; protection rate more than 70%; GMI more than 2.5 folds, the immunogenicity will reach the design requirements.

#### Statistics analysis of safety

After the first dose inoculation and the second dose inoculation, the number of adverse reactions (rate), number of cases and adverse reaction grade were recorded.

The number of adverse events after inoculation will be described.

Comparisons will be conducted to evaluate differences in response between study groups using a  $\chi^2$  test or Fisher's exact test to compare to the difference of adverse events rate. Statistical significance will be considered at a level of  $\alpha=0.05$  and all tests will be 2-sided.

#### Comparison of compliance

The rate of expulsion and the rate of drug combination will be described.

Comparisons will be conducted to evaluate differences in response between study groups using a  $\chi^2$  test or Fisher's exact test to compare to the difference of the rate of expulsion and the rate of drug combination. Statistical significance will be considered at a level of  $\alpha = 0.05$  and all tests will

be 2-sided.

## APPENDIX I. GRADING STANDARDS FOR SEVERITY OF SAFETY INFORMATION

The Event of clinical response and laboratory abnormalities after vaccination is judged by the China State Food and Drug Administration on "Guidelines for the classification of adverse events in vaccine clinical trials".

### **Grading of Local Adverse Events**

| Local Adverse Reactions | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe (Grade 3) | Potential Life Threatened (Grade 4) |
|---|---|---|---|---|
| Pain | Resistance or withdrawal after contact or touch | Crying after touching or touching, but soothing | There is no comfort in continual crying | Require emergency or hospitalization |
| Induration | Diameter < 2.5 cm | Diameter ≥2.5cm, and area < 50% of the inoculated limb (anatomically, the limb where the inoculated site is located, such as the upper arm or thigh) | Area ≥ 50% of inoculated limb<br>or ulceration or secondary<br>infection or phlebitis or wound<br>drainage | Abscesses, exfoliating dermatitis, and necrosis of the dermis or deep tissue |
| Redness | Diameter < 2.5 cm | Diameter ≥2.5cm, and area < 50% of the inoculated limb (anatomically, the limb where the inoculated site is located, such as the upper arm or thigh) | Area ≥ 50% of inoculated limb<br>or ulceration or secondary<br>infection or phlebitis or wound<br>drainage | Abscesses, exfoliating dermatitis, and necrosis of the dermis or deep tissue |

| Rash<br>Swelling | <15 mm and does not affect activity | 15-30 mm or affect activity | >30 mm or limit daily activity | Gangrene |
|---|---|---|---|---|
| Itching | 6 | The site of inoculation was itchy, which did not relieve within 48 | | N/A |
| 8 | 48 hours after treatment | hours after treatment | | |

## **Grading of Systemic Adverse Events**

| Systemic<br>Adverse<br>Reactions | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potential Life Threatened<br>(Grade 4) |
|---|---|---|---|---|
| Fever | 37.5-38.0°C | 38.0-39.5°C | ≥39.5°C | |
| Diarrhea | Mild or transient, $3 \sim 4$ stools per day or mild diarrhea lasting for less than 1 weeks | Moderate or persistent, 5~7 times per day, or more than 1 week diarrhea | > 7 times of water stool per day,<br>or blood diarrhea, orthostatic<br>hypotension | Hypotension shock requiring hospitalization |
| Constipation | Need stool softener and diet adjustment | Need a laxative | Stubborn constipation needs to be dredge manually or use enema | Toxic megacolon or ileus |
| Dysphagia | Slight discomfort in swallowing | Diet restricted | Diet and conversation are very limited; Cannot eat solid food | No liquid food; Need intravenous nutrition |
| Anorexia | Decreased appetite, but not reduced food intake | Decreased appetite, decreased food intake, but no significant weight loss | Decreased appetite and significantly decreased body weight | Need for intervention(E.g., gastric feeding, parenteral nutrition) |
| Vomiting | 1~2/24 hours with no impact on activities | 3~5/24 hours or restricted activities | >6 times within 24 hours or intravenous rehydration is required | Hospitalize or other routes of nutrition are required because of hypotensive shock. |

| Nausea Transient (<24 hours) or | | Reduced food intake due to | Persistent nausea causes almost | A threat to life(E.g. hypotensive |
|---|---|---|---|---|
| | intermittent and basically normal | persistent nausea (24~48 hours) | no food intake (>48 hours) or | shock) |
| | food intake | | requires intravenous fluids | |
| muscle pain | Do not affect daily activities | Slightly affect daily activities | Severe muscle pain that severely | Emergency or hospitalize |
| (Non- | | | affects daily activities | |
| inoculated | | | | |
| site) | | | | |
| Arthritis | Mild pain with inflammation, | Moderate pain with | Severe pain with inflammation, | Permanent and/or incapacitated |
| | erythema or joint swelling; But | inflammation, erythema or joint | erythema or joint swelling; | joint injury |
| | without hindrance to function | swelling; Hinder function, but do | Impact on daily activities | |
| | | not affect daily activities | | |
| Arthralgia | Mild pain, no impairment of | Moderate pain; Painkillers and/or | Severe pain; The need for | Impotence pain |
| | function | pain are required to interfere with | painkillers and/or pain affects | |
| | | function, but do not affect daily | daily activities | |
| | | activities | | |
| Headache | No effect on daily activities, no | Having a temporary effect on | Seriously affecting daily | Stubbornness, emergency or |
| | treatment required | daily activities and may require | activities, requiring treatment or | hospitalize |
| | | treatment or intervention. | intervention | |
| New | Duration of convulsions < 5 | Duration of convulsions ≥5~< | Duration of convulsions ≥ 20 | Prolonged and multiple |
| convulsions | minutes, and status after | 20 minutes, and status after | minutes or status after | convulsions (e.g., status |
| | convulsions <24 hours | convulsions <24 hours | convulsions >24 hours | |

| | T | | | 1 |
|---|---|---|---|---|
| | | | | convulsions) or difficult to |
| | | | | control (e.g., intractable epilepsy) |
| Cough | Transient, no treatment required | Keep coughing | Coughing, uncontrollable | Emergency or hospitalize |
| | | | treatment | |
| Difficulty in | Moving difficulty in breathing | Normal activity difficulty in | Rest time difficulty in breathing | Difficulty in breathing, need |
| breathing | | breathing | | oxygen therapy, hospitalize or |
| | | | | assisted breathing |
| Pruritus at | Slightly itchy, not affecting or | Itching affects everyday life | Pruritus makes daily life | NA |
| non-inoculated | slightly affecting everyday life | | impossible | |
| site (no skin | | | | |
| damage) | | | | |
| Abnormal | Erythema/pruritus/color Change | Diffuse rash/maculopapular | Blister/exudate/desquamate/ulcer | Exfoliative dermatitis involving |
| mucous | | rash/dry/detritus | | mucosa, or erythema multiforme, |
| membrane of | | | | or suspected Stevens-Johnsons |
| skin | | | | syndrome |
| Insomnia * | Mild difficulty in falling asleep, | Moderate difficulty in falling | Severe sleep difficulty, severe | NA |
| | not affecting or slightly affecting | asleep, affecting everyday life | impact on daily life, need to be | |
| | daily life | | treated or hospitalize | |
| To provoke or | Mild irritability or mild inhibition | Irritable or sleepy. | Unable to soothe or react poorly | NA |
| inhibit. | | | | |

| Acute allergic | Local urticaria (blister), no | Local urticaria, requiring | Extensive urticaria or | Anaphylactic shock or life- |
|---|---|---|---|---|
| reaction ** | treatment required | treatment or mild angioedema, no | angioedema requiring treatment | threatening bronchospasm or |
| | | treatment required | or mild bronchospasm | laryngeal edema |
| Fatigue, | Do not affect daily activities | Affect normal daily activities | Seriously affect daily activities, | Emergency or hospitalize |
| fatigue | | | unable to work | |
| Pain at non- | Mild pain, not affecting or | Pain affects everyday life | Pain does not work in everyday | Disabling pain, loss of basic self- |
| inoculated site | slightly affecting daily life | | life | care |
| #(Location | | | | |
| identified at | | | | |
| the time of | | | | |
| reporting) | | | | |

## **Grading of Blood Biochemical**

| Serum | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potential Life<br>Threatened<br>(Grade 4) |
|---|---|---|---|---|
| Elevated liver function caused by AST ALT, influence factors | 1.25-2.5 *ULN | 2.6-5*ULN | 5.1-10*ULN | >10*ULN |
| Creatinine | 1.1-1.5*ULN | 1.6-3.0*ULN | 3.1-6*ULN | >6*ULN |
| Urea nitrogen (BUN) | 1.25-2.5 *ULN | 2.6-5*ULN | 5.1-10*ULN | >10*ULN |
| Bilirubin: elevation caused by factors, but functional examination is normal | 1.1-1.5*ULN | 1.6-2.0*ULN | 2.0-3.0*ULN | >3.0*ULN |
| Bilirubin: the increase caused by the factors associated with the increase of liver function test index | 1.1-1.25*ULN | 1.26-1.5*ULN | 1.51-1.75*ULN | >1.75*ULN |

# **Grading of Blood Routine**

| Detection indicators | Level 1 | Level 2 | Level 3 | Level 4 |
|---|---|---|---|---|
| Liver function (ALT, AST increased) | 1. 25~<2. 5 ×ULN | 2.5~<5.0×ULN | 5.0~<10×ULN | ≥10×ULN |
| Total bilirubin increased (Mg/dL; Mmol/L) | 1. 1~<1. 6×ULN | 1.6~<2.6×ULN | 2.6~5.0×ULN | ≥5. 0×ULN |

# **Grading of Urine Routine**

| Test Indicators/Grades | Level 1 | Level 2 | Level 3 | Level 4 |
|---|---|---|---|---|
| WBC (109/L) | 11~<13 | 13~<15 | 15~<30 | ≥30 |
| WBC (109/L) | 2. 000 <sup>~</sup> 2. 499 | 1. 500 <sup>~</sup> 1. 999 | 1. 000 <sup>~</sup> 1. 499 | <1.000 |
| Lymphocyte Decrease (LY, 109/L) | 0. 75 <sup>~</sup> 1. 00 | 0. 5~0. 749 | 0. 25~0. 49 | <0. 25 |

| Neutropenia (ANC, 109/L) | 0.800~1.000 | 0. 600 <sup>~</sup> 0. 799 | 0. 400~0. 599 | <0.400 |
|---|---|---|---|---|
| Eosinophils (Eos, 109/L) | 0.65~1.5 | 1. 51~5. 0 | >5. 0 | High<br>eosinophil<br>syndrome |
| Thrombocytopenia (PLT, 109/L) | NA | 50 <sup>~</sup> 75 | 25 <sup>~</sup> 49 | <25 |
| Low hemoglobin (g/dL) | 9.5 <sup>~</sup> 10.4 | 8. 5 <sup>~</sup> <9. 5 | 6. 5 <sup>~</sup> <8. 5 | <6.5 |

# APPENDIX II. THE RELATIONSHIP BETWEEN ADVERSE EVENTS AND TRIAL VACCINES

**Absolutely unrelated**: Because of other factors lead to adverse events, there is evidence that adverse events are caused by other causes, not related to vaccination.

**Possible unrelated:** Adverse events probable be caused by other factors, such as the clinical status of the subjects, other treatment or concomitant medication, inconsistent with the known adverse reactions of vaccination.

**Quite possible related:** Adverse events are consistent with known information of vaccine, and there is a causal relationship with the vaccine, not by other factors, such as the clinical status of the subjects, or other treatment with medication.

**Possible related:** Adverse events are consistent with known information of vaccine, and there is a causal relationship with the vaccine, not by other factors, such as the clinical status of the subjects, or other treatment with medication.

**Related:** Adverse events are consistent with known information of vaccine, and there is a causal relationship with the vaccine, not by other factors, such as the clinical status of the subjects, or other treatment with medication. In addition, adverse events will be repeated when subjects are tested with the vaccine.